CLINICAL TRIAL: NCT05896358
Title: Dietary Treatment for Post Bariatric Weight Regain:Evaluation of the Efficacy of a KD
Brief Title: Dietary Treatment for Post Bariatric Weight Regain
Acronym: WRKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Full professor, University of Roma La Sapienza
Other Study IDs: 2023KDWR
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric naive: patients with obesity who have not undergone bariatric surgery in the past
  Interventions: Behavioral: ketogenic diet
- Post Bariatric: patients with obesity who have undergone bariatric surgery in the past and have experienced weight regain or insufficient weight loss
  Interventions: Behavioral: ketogenic diet

INTERVENTIONS:
Behavioral: ketogenic diet — a low calorie ketogenic diet

SUMMARY:
Metabolic surgery has, among all obesity treatments, the best long term efficacy, but weight regain (weight regain, WR) or insufficient weight loss (IWL) are relatively common. These are hard to treat, with dietary treatment often failing, and redo surgery being commonly proposed.The ketogenic diet is vastly utilised to obtain weight loss in obesity, but little data is available regarding its application on post bariatric patients. Ad hoc designed studies are needed to confirm the efficacy and safety of a VLCKD in the treatment of WR and IWL. The aim of this study is to test whether the ketogenic diet is a safe and effective treatment in post bariatric weight regain, compared to its application before bariatric surgery.

DETAILED DESCRIPTION:
Metabolic surgery is, to date, the strategy for the treatment of obesity with the greatest long-term efficacy. However, especially in those lost to surgical and nutritional follow-up, weight regain (weight regain, WR) or insufficient weight loss (IWL) are relatively common. In particular, depending on the type of surgery considered, it has been observed that up to 40% of subjects undergoing surgery report a WR long term, where data on IWL are still insufficient to draw well-defined estimates. WR and IWL are hard to treat, with dietary treatment often failing, and redo surgery being commonly proposed, with increased risk of complications and little effect.

The ketogenic diet is one of the pivotal dietary therapies for the treatment of obesity, with excellent evidence in terms of weight loss and improvement in complications of excess weight. Very little data is available regarding its application on post bariatric patients: Correa and colleagues reported in a retrospective case series the efficacy and safety of a very low calorie ketogenic diet (VLCKD) in 11 patients with IWL or WR after gastric bypass, reporting a good safety profile, good tolerability, and an average weight loss of 9 kg in 2 months of therapy. Although promising, the data in the literature are extremely scarce, and therefore ad hoc designed studies are needed to confirm the efficacy and safety of a VLCKD in the treatment of WR and IWL.

The objective of this study is to test whether the application of a ketogenic diet is a safe and effective treatment in post bariatric weight regain, compared to its application before bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

-obesity (BMI ≥ 30 Kg/m2)

Exclusion Criteria:

* Type 1 diabetes mellitus
* Renal failure (GFR<60)
* Liver failure (decompensated cirrhosis)
* Congenital metabolic diseases
* Pregnancy
* lactation
* Major psychiatric disorder
* Alcoholism
* drug addiction
* patients who are not self-sufficient and without adequate family and social support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre bariatric treatment arm will be composed of:
  -individuals with no history of bariatric surgery
  Post bariatric treatment arm will be composed of:
  * individuals with previous metabolic surgery (RYGB or Sleeve gastrectomy) and
  * excess WL < 50% at 18 months after surgery (IWL) or
  * clinically relevant WR after satisfactory WL
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
weight change | at baseline and right after the dietary intervention (8 weeks)
  body mass change (kg) within and between groups

SECONDARY OUTCOMES:
body fat change | at baseline and right after the dietary intervention (8 weeks)
  body fat change (kg) within and between groups
muscle mass change | at baseline and right after the dietary intervention (8 weeks)
  lean mass change (kg) within and between groups
waist circumference change | at baseline and right after the dietary intervention (8 weeks)
  waist circumference change (cm) within and between groups
mean blood pressure change | at baseline and right after the dietary intervention (8 weeks)
  mean blood pressure change (mmHg) within and between groups
glucose concentration change | at baseline and right after the dietary intervention (8 weeks)
  glucose change (mg/dL) within and between groups
insulin concentration change | at baseline and right after the dietary intervention (8 weeks)
  insulin change (UI/mL) within and between groups
uric acid concentration change | at baseline and right after the dietary intervention (8 weeks)
  uric acid change (mg/dL) within and between groups
creatinine concentration change | at baseline and right after the dietary intervention (8 weeks)
  creatinine change (mg/dL) within and between groups
cholesterol concentration change | at baseline and right after the dietary intervention (8 weeks)
  cholesterol change (mg/dL) within and between groups
triglycerides concentration change | at baseline and right after the dietary intervention (8 weeks)
  triglycerides change (mg/dL) within and between groups

CONTACTS AND LOCATIONS:
Overall Officials: lucio gnessi, Principal Investigator — sapienza università di roma
Locations (1):
- Sapienza University of Rome, Roma, Italy